CLINICAL TRIAL: NCT03384602
Title: Prevention of Cognitive Decline and Falls With Dalcroze Eurhythmics and a Simple Home Exercise Strength Program for Seniors With Subjective Cognitive Decline (SCD) - MOVE for Your MIND
Brief Title: MOVE for Your MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation, Switzerland (Unknown); University Hospital, Toulouse, France (Unknown); Waid City Hospital, Zurich, Switzerland (Unknown); Felix Platter Hospital, Basel, Switzerland (Unknown); JungDiagnostics, Hamburg, Germany (Unknown); Ferrari Data Solution (Other); Vontobel Foundation, Switzerland (Unknown); Age Stiftung, Zurich, Switzerland (Unknown); Gemeinnützige Stiftung EMPIRIS, Alzheimer Fund, Zurich Switzerland (Unknown); Stiftung für Demenzforschung in Basel, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-01288
Record Dates: First submitted 2017-10-16; First posted 2017-12-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Decline; Fall
Keywords: subjective cognitive decline; falls prevention; cognitive function; dalcroze eurhythmics; home exercise program; seniors
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Two intervention groups: Active I = Dalcroze Eurhythmic Program Active II: simple home exercise program Control group: no change in daily activities, no intervention
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dalcroze Eurhythmics program (Active Comparator): music-based multi-task exercise intervention
  Interventions: Other: Dalcroze Eurhythmics Program
- home exercise strength program (Active Comparator): simple strength training program to perform individually at home
  Interventions: Other: home exercise strength program
- Control group (No Intervention): no change in the daily activities, no exercise intervention

INTERVENTIONS:
Other: Dalcroze Eurhythmics Program — music-based multi-task exercise in group setting
  Arms: Dalcroze Eurhythmics program
Other: home exercise strength program — simple strength exercise program to perform individually at home
  Arms: home exercise strength program

SUMMARY:
Among the most promising interventions targeting both cognitive and functional decline, is Exercise. However, evidence regarding exercise interventions among seniors with cognitive impairment are inconclusive, likely due to challenges of recruitment and adherence. Alternatively, seniors with subjective cognitive decline (SCD), who are not yet meeting objective criteria of cognitive impairment, but have been shown to have twice the conversion rate to dementia compared with healthy seniors, are more likely to be motivated to participate and adhere to exercise interventions. Thus, exercise interventions in seniors with SCD may provide a window of opportunity for early prevention of dementia and falls.

The investigators aim to test the effect of a group exercise (multi-task Jaques-Dalcroze Eurhythmics) and a simple home strength exercise program on change of cognitive function and the rate of falling among seniors with SCD.

DETAILED DESCRIPTION:
In Europe and in Switzerland, the number of seniors age 70 and older is predicted to increase from 25% to 40% by 2030, as is the number of seniors with cognitive impairments, physical frailty and resulting consequences, such as falls and loss of autonomy. One out of three seniors age 65 and one out of two seniors age 80 experience at least one fall per year. Prevalence of dementia increases with age and more than doubles a seniors' risk of falling.

Among the most promising interventions targeting both cognitive and functional decline, is Exercise. However, evidence regarding exercise interventions among seniors with cognitive impairment are inconclusive, likely due to challenges of recruitment and adherence. Alternatively, seniors with subjective cognitive decline (SCD), who are not yet meeting objective criteria of cognitive impairment, but have been shown to have twice the conversion rate to dementia compared with healthy seniors, are more likely to be motivated to participate and adhere to exercise interventions. Thus, exercise interventions in seniors with SCD may provide a window of opportunity for early prevention of dementia and falls.

The investigators aim to test the effect of a group exercise (multi-task Jaques-Dalcroze Eurhythmics) and a simple home strength exercise program on change of cognitive function and the rate of falling among seniors with SCD.

The MOVE for your MIND trial will be a single center, single-blinded randomized controlled clinical trial among 195 senior men and women and a 12 month follow-up. Participants will be community-dwelling seniors, age 70+ who meet the criteria for SCD without evidence for objective cognitive impairment. The 3 treatment arms are: (1) Jaques-Dalcroze Eurhythmics group exercise (1x60min/week), (2) simple home exercise strength program (3x30min/week), (3) control group without exercise intervention. All participants will receive a monthly "Healthy Nutrition" lecture. The hypothesis is that both exercise groups are superior to control. Under these assumptions, and a sample size of 195 seniors, the investigators will have >90% power for change in cognitive function and >80% power for the difference in the rate of falls. Clinical visits will be at baseline, 6 months, and 12 months. Therapeutic interventions for seniors with early subjective signs of cognitive decline that are effective, affordable, and well-tolerated in the prevention of both, cognitive and physical function decline, are urgently needed and will have an outstanding impact on public health as a whole. To the investigator's knowledge, this is the first exercise trial to target seniors with SCD and with the change in cognitive function and the rate of falls as the primary endpoints. Providing an evidence-base for a group- and a home-based exercise will give a choice to patients. Further, the mechanistic biomarker study for brain and muscle health among seniors with SCD will support the findings at the cellular level and whole-brain MRI imaging will support them at a structural level.

ELIGIBILITY:
Inclusion Criteria:

* Age 70+, living in the community
* Meet the criterion for SCD defined by a score of ≥25 points on the MAC-Q questionnaire

Exclusion Criteria:

* Signs of mild cognitive impairment (MCI), MoCA score ≤24
* Score of ≥5 on the short form of the Geriatric Depression Scale (15items)
* Inability to walk or to come to the study entre
* Severe gait impairment or diseases with a risk of recurrent falling (e.g. Parkinson's disease/syndrome, Hemiplegia after stroke, symptomatic stenosis of the spinal canal, polyneuropathy, epilepsy, recurring vertigo, recurring syncope, heavy alcohol consumption)
* Currently engaged in regular (once a week or more) strength training instructed by a professional teacher and including the explicit aim to improve muscle strength, or regular (once a week or more) Dalcroze eurhythmics classes
* Active cancer or current cancer treatment
* Inability to read and/or speak German necessary to understand the instructions

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 195 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function | 12 months
  assessed with the CERAD-plus test
Rate of falls | 12 months
  The circumstances and injuries associated with the fall will be ascertained with a questionnaire.

SECONDARY OUTCOMES:
Proportion of seniors with any falls and injurious falls | 12 months
  Participants will record incident falls in the study diary.
Rate of injurious falls | 12 months
  The number of falls that resulted in any injury will be examined and categorized according to severity of the injury.
Cognitive function: verbal fluency test | 12 months
  The verbal fluency test (animal naming) is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Boston Naming test | 12 months
  The Boston Naming test (15 items) is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Mini Mental State Exam | 12 months
  The Mini Mental State Exam is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Word List Learning | 12 months
  Word List Learning is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Word List Recall | 12 months
  Word List Recall is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Word List Recognition | 12 months
  Word List Recognition (10 original words, 10 foils) is part of the CERAD-plus test battery (change over 12 months will be evaluated)
Cognitive function: Constructional Praxis | 12 months
  Constructional Praxis is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Constructional Praxis Recall | 12 months
  Constructional Praxis Recall is part of the CERAD test battery (change over 12 months will be evaluated)
Cognitive function: Trial Making Test A | 12 months
  The Trial Making Test A is part of the CERAD-Plus test battery (change over 12 months will be evaluated)
Cognitive function: Trial Making Test B | 12 months
  The Trial Making Test B is part of the CERAD-Plus test battery (change over 12 months will be evaluated)
Cognitive function: Phonematic Fluency Test | 12 months
  The Phonematic Fluency test (S-words) is part of the CERAD-Plus test battery (change over 12 months will be evaluated)
Incident MCI | 12 months
  Based on the results from the CERAD-plus test battery
Functional decline: gait speed | 12 months
  Gait speed will be measured with a stop watch over a distance of 4 meters.
Functional decline: timed up and go test | 12 months
  Assessed with the standard timed up and go test protocol
Functional decline: repeated sit-to-stand test | 12 months
  Assessed with the repeated sit-to-stand test protocol
Functional decline: grip strength | 12 months
  Assessed using a Martin Vigorimeter
Functional decline: short physical performance battery | 12 months
  Assessed using the short physical performance battery
Change in gait variability under single task condition | 12 months
  Assessed with a GAITRite® gait analysis system (Platinum CIR Systems, PA, USA) and/or Gait Up gait analysis system (Gait UP SA, Lausanne, Switzerland)
Change in gait variability under dual task condition | 12 months
  Assessed with a GAITRite® gait analysis system (Platinum CIR Systems, PA, USA) and/or Gait Up gait analysis system (Gait UP SA, Lausanne, Switzerland)
Quality of life: EuroQuol | 12 months
  Assessed using the German Version of EuroQuol EQ5D-3L questionnaire according to the Austrian reference scale
Quality of life: RAND 36-Item Short Form Survey | 12 months
  Assessed using the RAND 36-Item Short Form Survey (SF-36)
Mental Health: Geriatric Depression Scale | 12 months
  Assessed with the short form of the Geriatric Depression Scale (GDS)
Changes in IGF-1 | 12 months
  Blood marker analyses: IGF-1
Changes in biomarkers of inflammation: hr-CRP | 12 months
  Blood marker analyses: hr-CRP
Changes in biomarkers of inflammation: IL-6 | 12 months
  Blood marker analyses: IL-6

OTHER OUTCOMES:
Structural brain changes | 12 months
  Assessed by voxel based volumetry with a Siemens Avanto 1.5 T (Siemens Erlangen, Germany) deploying the classical dementia protocol (T2_tse_tra_512, T2_tirm_tra_dark-fl_5mm, T2_fl2d_tra_T2, T2_tse_cor_3mm, BC_t1_mpr_tra_iso_2, Ep2d_diff_tra). No contrast agents will be used.
Daily physical activity | 12 months
  assessed with the Nurse's Health Study physical activity questionnaire excerpt.
Effect of life-time physical activity | Baseline
  Retrospective Physical Activity Survey modified after Kriska et al. (1988)
TNF-alpha | 12 months
  Blood sample assessment: TNF-alpha
VEGF | 12 months
  Blood sample assessment: VEGF
BDNF | 12 months
  Blood sample assessment: BDNF
Sr IL-6 | 12 months
  Blood sample assessment: Sr IL-6
25-hydroxyvitamin D | 12 months
  Blood sample assessment: 25-hydroxyvitamin D
Hearing | 12 months
  Pure-tone testing in both ears
Effect of life-time cognitive activities | 12 months
  Cognitive Activities Questionnaire (CAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Heike A Bischoff, Prof. Dr. med., DrPH, Principal Investigator — University of Zurich
Locations (1):
- Centre on Aging and Mobility, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No